CLINICAL TRIAL: NCT06948253
Title: Comparing Postoperative Analgesic Techniques for Umbilical Hernia Repair: A Randomized Trial of Ultrasound Guided Caudal, Erector Spinae, and External Oblique Interfascial Plane Blocks
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Zakarea Wfa, Assisted professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 36264PR1119/3/25
Record Dates: First submitted 2025-04-17; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Regional Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group E (Active Comparator): Erector spinae plain block group will receive 0.5 ml/kg of 0.25%bupivacaine bilaterally
  Interventions: Other: External Oblique Intercostal Plane Block
- Group C (Active Comparator): Caudal block group will receive 1 ml/kg of 0.25% bupivacaine.
  Interventions: Other: Caudal Block Anesthesia
- Group EOI (Active Comparator): External oblique intercostal block will recive 0.5 ml/kg 0.25 % bupivacaine bilaterally.
  Interventions: Other: Erector Spinae Plane Block

INTERVENTIONS:
Other: Erector Spinae Plane Block — The correct location of the needle tip in the fascial plane deep to the erector spinae muscle will be conﬁrmed by injecting 0.5-1 ml of saline and observing the ﬂuid lifting the erector spinae muscle off the transverse process while avoiding muscle distension (hydro dissection)
  Arms: Group EOI
Other: Caudal Block Anesthesia — The needle will be advanced at a 20-degree angle with needle tip and length visualization. A pop can be appreciated as the needle passes through the sacrococcygeal ligament.
  Once the needle will be confirmed to be in the caudal space on the screen, carefully aspirate to confirm absence of CSF or blood.
  Arms: Group C
Other: External Oblique Intercostal Plane Block — the needle will be advanced until the tip lay in the plane between the external oblique muscle and intercostal muscles between the sixth and seventh ribs
  Arms: Group E

SUMMARY:
The aim of this study is to evaluate the efficacy of ultrasound guided Erector block versus caudal block versus external oblique intercostal plane block perioperatively

DETAILED DESCRIPTION:
umblical hernia repair surgeries have been performed in the practice of pediatric surgeries, ensuring adequate perioperative analgesia is crucial for perioperative care as pain in pediatric patients can cause functional recuperation and lead to negative behavioral changes and family dissatisfaction. (1) Various studies are made to improve postoperative analgesia and facilitate recovery in pediatric patients.(1) Day-case surgery is defined as the planned day admission of a patient to hospital for a surgical procedure, after which there is subsequent successful and safe discharge back home on the same day in a safe and timely manner instead of spending prolonged periods within the hospital.(2) This has significant implications, including reducing hospital stay, hospital-acquired infection, and healthcare-related costs while also improving patient experience and service efficiency. Surgical, anesthetic, and patient factors should be considered for successful day case surgery.(2) External oblique intercostal plane block (EOIPB) is a novel fascial plane block which aims to provide upper midline and lateral abdominal wall analgesia thereby reducing perioperative opioid consumption , LA is deposited into the fascial plane beneath the external oblique muscle (EOM) and superficial to the sixth rib or external intercostal muscle. It targets anterior and lateral cutaneous branches of the thoracoabdominal nerves from the ventral rami of spinal nerves.(3)

Caudal block is the most frequently performed regional technique for pain management in children undergoing lower abdominal surgeries. Ultrasound guidance has resulted in enhanced reliability and safety profiles for caudal blocks.(4) The erector spinae plane block (ESPB), multiple studies demonstrated its potential as a practical approach for managing postoperative pain in the last decade, involves an ultrasound-guided injection of a relatively large volume of local anesthetic into the fascial plane beneath the erector spinae muscle. (5)

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients of both sexes undergoing elective umblical hernia surgeries aged from 2 year to 7 years belonging to ASA I or II.

Exclusion Criteria:

* Parents refusal.
* Coagulopathy.
* Allergy to local anesthesia.
* Local infection at the site of injection.
* Neurological anomalies.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | 15 minute after operation , 30 minutes after operation and 4 h after operation
  Faces Legs Activity Cry Consolability tool (FLACC, 0- 10)

SECONDARY OUTCOMES:
Secondary outcome | 6 hours
  First dose of fentanyl as a rescue analgesia in dose of 0.5 μg/kg. Total doses of fentanyl as a rescue analgesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Zakarea Wfa, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided